CLINICAL TRIAL: NCT04704427
Title: Rehabilitative BCI for Lower Limb Function Recovery in Acute Ischemic Stroke
Brief Title: Rehabilitative BCI in Acute Ischemic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LYS[2020]-133
Record Dates: First submitted 2020-12-20; First posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-12

CONDITIONS: Stroke, Acute
Keywords: Brain Computer Interface; Lower Limb Function Recovery; Brain Machine Interface
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitative BCI training (Experimental): The experimental group will receive brain computer interface-based lower limb function training (BCI-LLT), 30 minutes/time, 5 times/week, with a 4-week training period.. The training using the lower limb orthosis targeted the patient's ability to walk.
  Interventions: Device: Non-invasive BCI training
- Traditional physical therapy protocol (Active Comparator): The control group will only receive traditional physical therapy protocol. The traditional physical therapy protocol of lower limb conducted with the same treatment frequency, intensity and duration of treatment, including muscle strength training, balance training and walking training, etc.
  Interventions: Other: Traditional Physiotherapy protocol

INTERVENTIONS:
Device: Non-invasive BCI training — In the experimental group, the participants receive non-invasive rehabilitative BCI training. The training using the lower limb orthosis targeted the patient's ability to walk.
  Arms: Rehabilitative BCI training
Other: Traditional Physiotherapy protocol — In the control group，the participants receive the traditional physiotherapy protocol, including muscle strength training, balance training and walking training, etc.
  Arms: Traditional physical therapy protocol

SUMMARY:
In order to explore the role and expound the mechanism of rehabilitative brain computer interface (BCI)-based training (referred to as the Walk Again Neurorehabilitation protocol) in neurofunctional reconstruction in acute phase of cerebral infarction, the investigators choose non-invasive BCI to study lower limb function of patients with acute cerebral infarction. The investigators evaluate lower limb function, the influence on the central brain functional network and relevant immuno-inflammatory indicators, so that the investigators can explore the therapeutic effect and mechanism in the acute phase of cerebral infarction and provide theoretical bases and feasible guidances for the treatment of post-stroke dyskinesia.

DETAILED DESCRIPTION:
The participants will be randomly divided into experimental group and control group. The experimental group will receive BCI-based lower limb functional training, 30 minutes per time, 5 times per week, with a 4-week training period; the control group will only receive routine lower limb training, with the same treatment frequency, intensity and duration. Statistical analysis will be performed to compare the relevant evaluation indexes of the experimental group and the control group after treatment and 90 days. In this study, the investigators will use Lower Extremity Fugl-Meyer Assessment (LE-FMA) to comprehensively evaluate the function of lower limbs, Functional Ambulation Category Scale (FAC) and 10-meter walking test (10MWT) for walking ability, modified Barthel index (MBI) for daily living abilities, functional magnetic resonance imaging（fMRI）and near infrared functional brain imaging (NIRS) to evaluate brain function and network reconstruction, the translocator protein(TSPO)-positron emission tomography (PET) and blood immune inflammation indicators to evaluate systemic and intracranial immune status.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of cerebral infarction conforms to the diagnostic criteria of "Chinese guidelines for diagnosis and treatment of acute ischemic stroke 2018".
2. 35 ≤ age ≤ 60 .
3. Onset (last-seen-well) time to randomization time from 24-72 hours.
4. First onset.
5. The lesion is assessed by MRI as a single subcortical infarction of the anterior circulation.
6. 5 ≤NIHSS≤15 (and 1 ≤6a/b≤3 ).
7. 1 ≤FAC functional walking scale score ≤ 3.
8. Signed informed consent from subject or legally authorized representative.

Exclusion Criteria:

1. Unstable vital signs.
2. Progressive stroke.
3. Patients have received intravenous thrombolysis or endovascular treatment.
4. Cardiogenic cerebral embolism.
5. Presence of moderate or higher vascular stenosis or vulnerable plaque based on Imaging assessment.
6. With other diseases of the nervous system.
7. With serious diseases of other systems (severe circulatory system, respiratory system, motor system) and other diseases unsuitable for training, such as atrial fibrillation, heart failure, lung infection, severe liver or kidney insufficiency, lower extremity venous thrombosis.
8. Lower limb dysfunction caused by other reasons, such as fracture, lower limb deformity, etc.
9. With contraindications in imaging examinations, such as metal implantation, fear of claustrophobia, and severe obesity.
10. Patient who cannot cooperate with training, such as mental disorders, cognitive dysfunction, Mini-Mental State Examination (MMSE) <21 points, etc.
11. Other reasons: alcoholism; pregnancy; skull defect; indwelling urinary catheter; vision defects affect training, etc.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-16 (Estimated); Primary Completion 2021-12-25 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Fugl-Meyer score of lower limbs from baseline to 4 weeks. | 0-4 weeks.
  It consists of 17 individual assessments that are summed to generate a total score. Scores range from 0-34, the higher the better.

SECONDARY OUTCOMES:
Functional ambulation category scale | 4 weeks and 90 days.
  This scale indicates the ability to walk independently and serves as the primary outcome measure.Participants will be asked to walk at their normal comfortable pace (handheld assistive device is acceptable if needed).
10-meter walk test | 4 weeks and 90 days.
  Gait speed will be measured as the average of 3 times 10-meter walk tests. Participants will be asked to walk at their normal comfortable pace (handheld assistive device is acceptable if needed).
Modified Barthel index | 4 weeks and 90 days.
  Scale range: 0-100 (with higher scores indicating a greater ability to complete activities of daily living)
National Institutes of Health Stroke Scale | 4 weeks and 90 days.
  The National Institutes of Health Stroke Scale (NIHSS) is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. The range of scores is from 0 (normal) to 42, with higher scores indicating greater stroke severity.
Gait analysis ( stride frequency, step length and velocity) | 4 weeks and 90 days.
  To evaluate the walking ability
Nodal functional connectivity strength analysis by functional magnetic resonance imaging | 4 weeks and 90 days.
  To evaluate the brain function and network
Changes in oxyhaemoglobin in related cortex by Functional near-infrared spectroscopy | 4 weeks and 90 days.
  To evaluate the brain cortex function.
The translocator protein(TSPO)-positron emission tomography (PET) | 4 weeks.
  Respond to inflammation in the brain
Fugl-Meyer score of lower limbs | 90 days.
  It consists of 17 individual assessments that are summed to generate a total score. Scores range from 0-34, the higher the better.

CONTACTS AND LOCATIONS:
Overall Officials: Guoguang Zhao, Principal Investigator — Xuanwu Hospital, Beijing

REFERENCES:
- [Background] Jackson A, Zimmermann JB. Neural interfaces for the brain and spinal cord--restoring motor function. Nat Rev Neurol. 2012 Dec;8(12):690-9. doi: 10.1038/nrneurol.2012.219. Epub 2012 Nov 13. PMID 23147846
- [Background] Ramos-Murguialday A, Broetz D, Rea M, Laer L, Yilmaz O, Brasil FL, Liberati G, Curado MR, Garcia-Cossio E, Vyziotis A, Cho W, Agostini M, Soares E, Soekadar S, Caria A, Cohen LG, Birbaumer N. Brain-machine interface in chronic stroke rehabilitation: a controlled study. Ann Neurol. 2013 Jul;74(1):100-8. doi: 10.1002/ana.23879. Epub 2013 Aug 7. PMID 23494615
- [Background] Lopez-Larraz E, Sarasola-Sanz A, Irastorza-Landa N, Birbaumer N, Ramos-Murguialday A. Brain-machine interfaces for rehabilitation in stroke: A review. NeuroRehabilitation. 2018;43(1):77-97. doi: 10.3233/NRE-172394. PMID 30056435
- [Background] Chaudhary U, Birbaumer N, Ramos-Murguialday A. Brain-computer interfaces for communication and rehabilitation. Nat Rev Neurol. 2016 Sep;12(9):513-25. doi: 10.1038/nrneurol.2016.113. Epub 2016 Aug 19. PMID 27539560
- [Background] Lebedev MA, Nicolelis MA. Brain-Machine Interfaces: From Basic Science to Neuroprostheses and Neurorehabilitation. Physiol Rev. 2017 Apr;97(2):767-837. doi: 10.1152/physrev.00027.2016. PMID 28275048
- [Background] Donati AR, Shokur S, Morya E, Campos DS, Moioli RC, Gitti CM, Augusto PB, Tripodi S, Pires CG, Pereira GA, Brasil FL, Gallo S, Lin AA, Takigami AK, Aratanha MA, Joshi S, Bleuler H, Cheng G, Rudolph A, Nicolelis MA. Long-Term Training with a Brain-Machine Interface-Based Gait Protocol Induces Partial Neurological Recovery in Paraplegic Patients. Sci Rep. 2016 Aug 11;6:30383. doi: 10.1038/srep30383. PMID 27513629
- [Background] Selfslagh A, Shokur S, Campos DSF, Donati ARC, Almeida S, Yamauti SY, Coelho DB, Bouri M, Nicolelis MAL. Non-invasive, Brain-controlled Functional Electrical Stimulation for Locomotion Rehabilitation in Individuals with Paraplegia. Sci Rep. 2019 May 1;9(1):6782. doi: 10.1038/s41598-019-43041-9. PMID 31043637